CLINICAL TRIAL: NCT00863369
Title: A Phase I/II Study of VELCADE in Combination With Gemcitabine in Relapsed B-Cell Non-Hodgkin's Lymphoma
Brief Title: Bortezomib and Gemcitabine in Treating Patients With Relapsed B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04115; P30CA033572 (NIH); CHNMC-04115; MILLENNIUM-CHNMC-04115; CDR0000637492 (Registry Identifier: NCI PDQ); NCI-2010-00925 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2023-03

CONDITIONS: Lymphoma
Keywords: recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; adult grade III lymphomatoid granulomatosis
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Rituximab; Bortezomib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bortezomib, gemcitabine hydrochloride, rituximab) (Experimental): Patients receive bortezomib IV, gemcitabine hydrochloride IV over 3-4 hours, and rituximab IV on days 1 and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: bortezomib; Drug: gemcitabine hydrochloride; Other: questionnaire administration

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Other: questionnaire administration — Ancillary studies

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with gemcitabine hydrochloride and rituximab may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of bortezomib and gemcitabine hydrochloride when given together with rituximab and to see how well they work in treating patients with progressive or relapsed B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary:

I. To evaluate the safety and feasibility of combining VELCADE (bortezomib) with gemcitabine (gemcitabine hydrochloride) in patients with recurrent lymphoma after standard therapy.

II. To define the maximum tolerated dose (MTD) of gemcitabine and Rituxan (rituximab) administered in combination with VELCADE given on a 21-day (old schema - Schema I) or 28-day (amended schema - Schema II) schedule.

Secondary:

I. To obtain preliminary data for response to this regimen in this patient population.

OUTLINE: This is a phase I, dose-escalation study of bortezomib and gemcitabine hydrochloride followed by a phase II study.

Patients receive bortezomib intravenously (IV), gemcitabine hydrochloride IV over 3-4 hours, and rituximab IV on days 1 and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed intermediate or high grade B-cell Non-Hodgkin lymphoma with primary progressive or relapsed disease
* Patients may have had up to 4 prior chemo-and-or radiation therapy regiments, including one autologous transplant based protocol; any prior therapy (chemotherapy or radiation) must have been completed at least 4 weeks prior to start of this protocol; for prior high-dose chemotherapy with stem cell transplant, a 6-week interval is required; all side effects must have resolved
* Karnofsky performance status >= 60%
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,500 mm^3
* Platelets >= 50,000 mm^3
* Total bilirubin =< 1.5 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min for creatinine levels above institutional normal (calculated or measured)
* Cardiac ejection fraction of > 40% by echocardiogram or multi gated acquisition (MUGA) scan
* Have no serious or intercurrent medical illness
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Patient has a platelet count of < 20 x 10^9/L with 7 days before enrollment
* Patient has an absolute neutrophil count of < 1.0 x 10^9/L within 7 days before enrollment
* Patient has a calculated or measured creatinine clearance of < 30 ml/min with 14 days before enrollment
* Patient has >= Grade 2 peripheral neuropathy within 14 days before enrollment
* Patient has hypersensitivity to bortezomib, boron, or mannitol
* Female subject is pregnant or breastfeeding; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for postmenopausal or surgically sterilized women
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patients who have had more than 4 prior different chemotherapy regimens will be excluded; patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for autologous transplant regimens) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not have previously received VELCADE or gemcitabine
* Patients with active central nervous system (CNS) involvement are not eligible
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-06-29 (Actual); Primary Completion 2016-08-25 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Popplewell, MD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2: Patients receive 1.0 mg/m2 of velcade IV days 1, 4, 8, 11, and 1000 mg/m2 of gemcitabine hydrochloride IV over 3-4 hours. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
- Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2: Patients receive 1.0 mg/m2 of velcade IV days 1, 4, 8, 11, and 800 mg/m2 of gemcitabine hydrochloride IV over 3-4 hours. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
- Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2: Patients receive 1.0 mg/m2 of velcade IV days 1, 15, and 800 mg/m2 of gemcitabine hydrochloride IV over 3-4 hours. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
- Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2: Patients receive 1.3 mg/m2 of velcade IV days 1, 15, and 800 mg/m2 of gemcitabine hydrochloride IV over 3-4 hours. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
- Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2: Patients receive 1.3 mg/m2 of velcade IV days 1, 15, and 1000 mg/m2 of gemcitabine hydrochloride IV over 3-4 hours. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
- Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2: Patients receive 1.3 mg/m2 of velcade IV days 1, 15, and 800 mg/m2 of gemcitabine hydrochloride IV over 3-4 hours 375 mg/m2 of rituximab IV on days 1 and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2
Started | 4 | 5 | 4 | 3 | 6 | 11
Completed | 4 | 5 | 4 | 3 | 6 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2 | Total
Number analyzed (Participants) | 4 | 5 | 4 | 3 | 6 | 11 | 33
Age, Continuous [Median (Full Range); unit: years] | 60 [55 to 67] | 50 [34 to 69] | 58 [41 to 66] | 66 [60 to 69] | 72 [58 to 77] | 66 [29 to 77] | 65 [29 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 0 | 2 | 4 | 10
  Male | 1 | 4 | 4 | 3 | 4 | 7 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1 | 3 | 0 | 5
  Hispanic | 1 | 0 | 1 | 0 | 0 | 2 | 4
  White Non-Hispanic | 3 | 4 | 2 | 2 | 3 | 8 | 22
  Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 4 | 3 | 6 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Dose Limiting Toxicity (DLT)
Description: Adverse events were graded by NCI CTCAE, Version 3.0. DLT defined as grade 4 thrombocytopenia, or grade 3 thrombocytopenia lasting greater than 7 days. Grade 4 neutropenia lasting 7 days or more despite use of growth factors. Febrile neutropenia only is it occurs after 7 days of neutropenia. Any grade 3 or higher non-hematologic toxicity related to the study drug, with the exception of alopecia, inadequately treated nausea, vomiting and/or diarrhea and fatigue.
Time Frame: 28 days from start of treatment, up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2
Number analyzed (Participants) | 4 | 5 | 4 | 3 | 6 | 11
Participants | 3 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Recommended Phase II Dose
Description: The maximum tolerated dose (MTD) of Gemcitabine in combination with 1.3 mg/m2 of velcade on days 1 and 15 is based on toxicities observed during the first cycle and is defined as the highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. Dose escalations proceeded according to a standard 3+3 design.
Time Frame: 28 days from start of treatment, up to 2 years.
Measure: Number; unit: mg/m^2
Groups:
- Treatment (Velcade, Gemcitabine Hydrochloride, Rituximab): Patients start with a dose of 1.0 mg/m2 velcade and 800 mg/m2 gemcitabine hydrochloride IV on days 1 and 8. Schedule of velcade\gemcitabine modified to days 1 and 15 with addition of 375 mg/m2 of rituximab on days 1 and 15. Treatment repeats every 28 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
  bortezomib: Given IV
  gemcitabine hydrochloride: Given IV
Arm/Group | Treatment (Velcade, Gemcitabine Hydrochloride, Rituximab)
Number analyzed (Participants) | 11
mg/m^2 | 1000

3. Secondary Outcome: Number of Subject With Complete Response
Description: Per standard lymphoma response criteria (Cheson): Complete Response (CR), 1. Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease related symptoms if present before therapy, with normalization of LDH if elevated prior to therapy. 2. All lymph nodes and masses must regress to normal size (<1.5 cm in greatest transverse diameter if >1.5 cm prior to treatment). 3. The spleen, if enlarged prior to therapy, must have regressed to normal size. 3. If bone marrow was involved by lymphoma, it must be cleared as documented by biopsy at the same location.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2
Number analyzed (Participants) | 4 | 5 | 4 | 3 | 6 | 11
Participants | 1 | 0 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 3 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2 | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2
All-Cause Mortality (participants affected / at risk) | 3/4 | 4/5 | 4/4 | 3/3 | 4/6 | 10/11
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/5 | 3/4 | 0/3 | 0/6 | 4/11
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 4/4 | 3/3 | 6/6 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2 (N=4) | Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 (N=5) | Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 (N=4) | Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2 (N=3) | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2 (N=6) | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2 (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets (Investigations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 Tx Schema I - Velcade 1.0 mg/m2, Gemcitabine 1000 mg/m2 (N=4) | Dose Level Tx Schema I -1 - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 (N=5) | Dose Level 3B Tx Schema II - Velcade 1.0 mg/m2, Gemcitabine 800 mg/m2 (N=4) | Dose Level 4B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 800 mg/m2 (N=3) | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2 (N=6) | Dose Level 5B Tx Schema II - Velcade 1.3 mg/m2, Gemcitabine 1000 mg/m2, Rituximab 375 mg/m2 (N=11)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 3 (14) | 5 (15) | 3 (10) | 1 (2) | 6 (26) | 10 (33)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (5) | 2 (2) | 2 (3) | 0 (0) | 3 (5) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (2) | 1 (2) | 2 (5) | 1 (2)
Distension/bloating, abdominal (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 4 (8)
Obstruction, GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Constitutional Symptoms - Other (Specify, __) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death not associated with CTCAE term (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema:limb (General disorders) | 1 (7) | 1 (3) | 0 (0) | 0 (0) | 2 (6) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (7) | 5 (13) | 2 (8) | 1 (2) | 2 (2) | 6 (16)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Flu-like syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Injection site reaction/extravasation changes (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - Other (Specify, __) (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Viral hepatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prolonged chest tube drainage or air leak after pulmonary resection (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication, non-infectious (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AGC (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 4 (10) | 5 (10) | 4 (13) | 2 (4) | 2 (5) | 6 (9)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 (5) | 5 (9) | 3 (9) | 2 (4) | 1 (5) | 6 (7)
Alkaline phosphatase (Investigations) | 1 (2) | 2 (4) | 3 (8) | 1 (2) | 0 (0) | 4 (5)
Bilirubin (hyperbilirubinemia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coagulation - Other (Specify, __) (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 1 (2) | 2 (4) | 3 (9) | 0 (0) | 1 (2) | 2 (3)
FEV(1) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytes (total WBC) (Investigations) | 3 (13) | 5 (13) | 2 (2) | 2 (3) | 4 (5) | 9 (34)
Lymphopenia (Investigations) | 3 (14) | 4 (12) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic/Laboratory - Other (Specify, __) (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 (8) | 5 (7) | 2 (2) | 2 (3) | 3 (4) | 8 (29)
Platelets (Investigations) | 3 (12) | 5 (15) | 3 (5) | 3 (7) | 4 (12) | 7 (27)
Vital capacity (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1)
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (8) | 5 (12) | 2 (9) | 2 (3) | 2 (4) | 5 (8)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (6) | 1 (1) | 2 (2) | 3 (6)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 4 (15)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 2 (6) | 0 (0) | 3 (6) | 2 (3)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (7) | 1 (1)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (3) | 1 (1) | 3 (7) | 2 (2)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 1 (3) | 0 (0) | 3 (3) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (4)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 2 (4) | 2 (3) | 2 (3) | 5 (8)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (3) | 1 (1) | 1 (3) | 0 (0) | 1 (2) | 2 (4)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 3 (6)
Pain (Musculoskeletal and connective tissue disorders) | 2 (9) | 4 (8) | 3 (9) | 0 (0) | 2 (4) | 9 (34)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 3 (11) | 3 (5) | 2 (2) | 1 (3) | 2 (9) | 5 (14)
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Taste alteration (dysgeusia) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Mood alteration (Psychiatric disorders) | 1 (2) | 4 (10) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (5) | 4 (6)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (4)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Pulmonary fibrosis (radiographic changes) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Induration/fibrosis (skin and subcutaneous tissue) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular - Other (Specify, __) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes